CLINICAL TRIAL: NCT03589794
Title: A Phase I Challenge Study to Evaluate Safety, Immunogenicity, and Efficacy of a Malaria Vaccine (rCSP Adjuvanted With AP 10-602 [GLA-LSQ]), in Healthy Adults
Brief Title: rCSP/AP10-602 [GLA-LSQ] Vaccine Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 13-0088; HHSN272201300022I
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2021-04-19

CONDITIONS: Plasmodium Falciparum Infection
Keywords: AP 10-602 [GLA-LSQ]; Challenge; Healthy adults; Malaria; P. falciparum; rCSP; Vaccine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1 (Experimental): 10 subjects receive 10 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ) intramuscularly (IM) on days 1, 29 and 85.
  Interventions: Other: AP10-602; Biological: rCSP
- Group 2 (Experimental): 10 subjects receive 30 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ) intramuscularly (IM) on days 1, 29 and 85.
  Interventions: Other: AP10-602; Biological: rCSP
- Group 3 (Experimental): 10 subjects receive 30 mcg rCSP intramuscularly (IM) on days 1, 29 and 85.
  Interventions: Biological: rCSP
- Group 4 (Experimental): 9 subjects receive 60 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ) intramuscularly (IM) on days 1 and 85. Subjects will then receive CHMI challenge with P. falciparum parasites of the NF54/3D7 strain on day 113.
  Interventions: Other: AP10-602; Other: Malaria challenge; Biological: rCSP
- Group 4B (Experimental): 10 subjects receive 60 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ) intramuscularly (IM) on days 1, 29 and 85. Subjects will then receive CHMI challenge with P. falciparum parasites of the NF54/3D7 strain on day 113.
  Interventions: Other: AP10-602; Other: Malaria challenge; Biological: rCSP
- Group 5 (Experimental): 10 subjects receive 10 mcg or 30 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ) intramuscularly (IM) on days 1, 29 and 85 if immunogenicity analysis conducted 28 days post-2nd dose in Groups 1, 2, and 3 show promise (at least fourfold increase in geometric mean anti-CSP antibody or geometric mean anti-CSP titer of 20). Otherwise, subjects will receive 60 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ). Subjects will then receive CHMI challenge with P. falciparum parasites of the NF54/3D7 strain on day 113.
  Interventions: Other: AP10-602; Other: Malaria challenge; Biological: rCSP
- Group 6 (Other): 6 subjects receive CHMI challenge with P. falciparum parasites of the NF54/3D7 strain.
  Interventions: Other: Malaria challenge

INTERVENTIONS:
Other: AP10-602 — Glucopyranosyl Lipid A -liposome-Quillaja Saponaria 21 (GLA-LSQ).
  Arms: Group 1; Group 2; Group 4; Group 4B; Group 5
Other: Malaria challenge — Exposure to mosquitoes infected with P. falciparum.
  Arms: Group 4; Group 4B; Group 5; Group 6
Biological: rCSP — The rCSP malaria vaccine is a recombinant full-length P. falciparum circumsporozoite protein comprised of an amino terminus that binds heparin-sulfate proteoglycans, a four-amino-acid repeat region and a carboxy-terminus that contains a thrombospondin-like Type I region domain.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 4B; Group 5

SUMMARY:
This is a study to evaluate the safety, immunogenicity, and efficacy of a recombinant circumsporozoite protein (rCSP) malaria vaccine administered with and without AP 10-602 [Glucopyranosyl Lipid A (GLA) in liposome Quillaja saponaria 21 formulation (LSQ)] adjuvant. 59 healthy adult, malaria naive volunteers aged 18 to 45 will receive vaccination with or without adjuvant (10 of those volunteers will receive rCSP alone) in five dose escalating groups. Each group will receive 3 vaccination doses total, with intramuscular (IM) injections on days 1, 29, and 85. A sixth group of 6 volunteers will receive no vaccinations and will participate as a control in a Controlled Human Malaria Infection (CHMI) challenge with two of the vaccinated groups. The study will be conducted at the Center for Vaccine Development (CVD) in Baltimore, Maryland. The patient participation duration is expected to be up to 886 days (up to 117 days for nonvaccination group). This study will test two hypotheses: (1) the rCSP/AP 10-602 [GLA-LSQ] candidate malaria vaccine will induce an immune response in a dose-dependent manner as measured by anti-CSP antibody titer via ELISA and (2) the rCSP/AP 10-602 [GLA-LSQ] candidate malaria vaccine will provide a minimum of 50% efficacy in vaccines compared to unvaccinated infectivity controls. The primary objective is to assess the safety and reactogenicity of candidate rCSP/AP 10-602 [GLA-LSQ] malaria vaccine when administered intramuscularly on a 1, 29, and 85 day schedule (Groups 1-3, 4B, 5) and on a 1 and 490 day schedule (Group 4) to healthy malaria-naive adults aged 18-45 years.

DETAILED DESCRIPTION:
This is a phase I, single-site, dose escalation study to evaluate the safety, immunogenicity, and efficacy of the recombinant circumsporozoite protein (rCSP) antigen malaria vaccine administered with and without AP 10-602 [Glucopyranosyl Lipid A (GLA) in liposome Quillaja saponaria 21 formulation (LSQ)]. The study population will consist of 65 healthy male and female adults aged 18 to 45 years old and be conducted at the Center for Vaccine Development (CVD) in Baltimore, Maryland. 49 healthy, malaria-naïve volunteers will receive rCSP vaccination with AP 10-602 [GLA-LSQ] adjuvant. Ten volunteers will receive rCSP alone. Each dose-escalating group will receive 3 intramuscular (IM) total doses of vaccine on days 1, 29, and 85. Group 1 will receive a dose of 10 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ) at each injection; Group 2 will receive 30 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ); Group 3 will receive 30 mcg rCSP without adjuvant; and Group 4 will receive 60 mcg rCSP + AP 10-602 [GLA-LSQ] (5 mcg GLA - 2 mcg LSQ). The dose for Group 5 will depend on immunogenicity analysis from groups 1, 2 and 3. If immunogenicity analysis conducted 28 days post-2nd dose in Groups 1, 2 and 3 show promise (at least fourfold increase in geometric mean anti-CSP antibody or geometric mean anti-CSP titer of 20), the 10 volunteers in Group 5 will receive the lowest rCSP dose that gives this predefined immunogenic response ((either 10 or 30 mcg rCSP) + AP 10-602 [GLA-LSQ],]), otherwise, Group 5 will receive 60 mcg rCSP + AP 10-602 [GLA-LSQ]. Groups will be vaccinated in a stepwise manner following a "telescoped" design. A sixth group of 6 volunteers (Group 6) will receive no vaccinations and will be used as an infectivity control for a Controlled Human Malaria Infection (CHMI) challenge. Groups 4 and 5 will also undergo the CHMI challenge together, 28 days after the last vaccination. The patient participation duration is expected to be up to 886 days for Groups 1, 2, 3, 4, and 5; and up to 117 days for Group 6. This study will test two hypotheses: (1) the rCSP/AP 10-602 [GLA-LSQ] candidate malaria vaccine will induce an immune response in a dose-dependent manner as measured by anti-CSP antibody titer via ELISA and (2) the rCSP/AP 10-602 [GLA-LSQ] candidate malaria vaccine will provide a minimum of 50% efficacy in vaccines compared to unvaccinated infectivity controls. The primary objective is to assess the safety and reactogenicity of candidate rCSP/AP 10-602 [GLA-LSQ] malaria vaccine when administered intramuscularly on a 1, 29, and 85 day schedule (Groups 1-3, 4B, 5) and on a 1 and 461 day schedule (Group 4) to healthy malaria-naive adults aged 18-45 years. The secondary objectives are to (1) assess immunogenicity of rCSP/AP 10-602 [GLA-LSQ] malaria vaccine when administered intramuscularly on a 1, 29, and 85 day (Groups 1-3, 4B, 5) and on a 1 and 490 day schedule (Group 4) schedule and (2) to assess the preliminary efficacy of candidate rCSP/AP 10-602 [GLA-LSQ] malaria vaccine against infection with Plasmodium falciparum malaria (defined as P. falciparum asexual parasitemia or a delay in patency of infection > 2 days versus unimmunized infectivity controls) under Controlled Human Malaria Infection (CHMI).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (males and non-pregnant, non-lactating females) between the ages of 18 and 45 years, inclusive
2. Able and willing to participate for the duration of the study
3. Able and willing to provide written (not proxy) informed consent
4. Provides informed consent and correctly answers > / = 70 percent on the post consent quiz before any study procedures and is available for all study visits
5. Females of childbearing potential and males must agree to practice highly effective contraception*

   *Contraception must be practiced from 30 days before the time of enrollment until at least 30 days following the third vaccine dose for groups 1, 2 and 3, and the malaria challenge event for groups 4, 4B, 5 and 6 (such as double barrier methods (condoms plus foam or spermicide, diaphragm plus foam or spermicide), licensed intrauterine devices (IUDs), intravaginal or intra/transdermal or oral hormonal methods initiated at least 30 days before inoculation or challenge, documented surgical sterilization via tubal ligation the essure procedure or hysterectomy, abstinence or a vasectomized partner). The contraceptive method should remain unchanged throughout the study participation
6. Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature); medical history; laboratory values* that do not meet toxicity grading criteria, except when Grade 1 and clinically insignificant; and a physical examination

   *Laboratory values include: hemoglobin, white blood cell count, platelet count, glucose (random), serum alanine aminotransferase (ALT), serum creatinine, urine protein and urine blood
7. Agree not to travel to a malaria endemic region during the entire course of the trial
8. Willing to avoid non-study related blood donation for the duration of participation in the study or until at least 1 year after receiving the last investigational vaccine, whichever is longer
9. Able to understand and comply with planned study procedures including daily outpatient follow-up visits beginning 5 days after malaria challenge (groups 4, 4B, 5 and 6 only)
10. Willing to avoid non-study related blood donation for 3 years following P. falciparum challenge (groups 4, 4B, 5 and 6 only)

Exclusion Criteria:

1. Any history of malaria infection, or travel to a malaria endemic region within 6 months before first vaccination
2. History of long-term residence (> / = 5 years) in an area known to have significant transmission of P. falciparum
3. Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg)
4. Positive sickle cell screening test or known hemoglobinopathy (groups 4, 4B, 5 and 6 only)
5. Current or recent (within the last four weeks) treatment with parenteral or oral corticosteroids (intranasal or inhaled steroids are acceptable), or other immunosuppressive agents, or chemotherapy
6. History of splenectomy
7. Participants who have a clinically significant (as determined by the PI or designee) baseline Grade 1 or greater toxicity, or any Grade 2 or greater toxicity (regardless of clinical significance) by the toxicity table, except hematuria > 1+ detected during menses for females*

   * For females who are menstruating, urinalysis frequently tests positive for blood and is not an indicator of poor health status or increased risk.
8. Vaccination with a live vaccine within the past 30 days or with a nonreplicating, inactivated, or subunit vaccine within the last 14 days
9. Known hypersensitivity to components of the vaccine for groups 1, 2, 3, 4, 4B and 5; or to the adjuvant for groups 1, 2, 4, 4B and 5
10. History of acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, nervous system, or other metabolic or autoimmune/inflammatory conditions
11. History of anaphylaxis or severe hypersensitivity reaction
12. History of Guillain-Barre syndrome or severe adverse reaction to any vaccination
13. Severe asthma, as defined by an emergency room visit or hospitalization within the last 12 months
14. Pregnant or breastfeeding women or women who plan to become pregnant before day 115 in groups 1, 2 and 3; or before 30 days post-malaria challenge in groups 4, 4B, 5 and 6
15. Concurrent participation in other investigational protocols prior to Day 141 or receipt of an investigational product within the previous 30 days
16. Planned receipt of an investigational product within 28 days following the last vaccination dose or malaria challenge
17. Any condition that, in the opinion of the investigator, would affect a participant's ability to understand or comply with the study protocol or would jeopardize a participant's safety or rights
18. History of previous receipt of a candidate malaria vaccine or a vaccine containing the GLA-LSQ adjuvant
19. Use or planned use of any drug with anti-malarial* activity 30 days before, or after malaria challenge (groups 4, 4B, 5 and 6 only)

    *Medications with antimalarial activity include trimethoprim-sulfamethoxazole, azithromycin, erythromycin, tetracycline, doxycycline, minocycline, clindamycin, ciprofloxacin, levofloxacin, norfloxacin and rifampin
20. Planned surgery 30 days before or after vaccination or malaria challenge
21. History of drug or alcohol abuse within the last five years
22. Receipt of blood or blood products in the previous six months or donation of a unit of blood within two months before screening
23. History of schizophrenia, bipolar disorder or other psychiatric condition that makes study compliance difficult*

    * Subjects with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide
24. History of diabetes mellitus with the exception of pregnancy-induced diabetes that has resolved
25. Has evidence of increased cardiovascular disease risk* (defined as > 10 percent, 5 year risk) as determined by the method of Gaziano (groups 4, 4B, 5 and 6 only)

    * Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg / mm^2), reported diabetes status, and blood pressure
26. Abnormal screening ECG* (groups 4, 4B, 5, and 6 only)

    * Pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial or ventricular contractions, right of left bundle branch block, advanced A-V heart block (secondary or tertiary), QT/QTc interval > 450 ms
27. Known hypersensitivity to mosquito bites, artemether-lumefantrine or atovaquone-proguanil (groups 4, 4B, 5 and 6 only)
28. Anticipated medication use during the 28-day post-challenge period that are known to interact with artemether/lumefantrine or atovaquone/proguanil, such as cimetidine, metoclopramide, antacids, and kaolin (groups 4, 4B, 5 and 6 only)
29. Previous participation in a CHMI study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting Adverse Events of Special Interest (AESIs) | Day 1 to Day 450
  According to the Medical Dictionary for Regulatory Activities (MedDRA) classification
Number of subjects reporting serious adverse events (SAEs) | Day 1 to Day 450
  According to the Medical Dictionary for Regulatory Activities (MedDRA) classification
Number of subjects reporting serious adverse events (SAEs) considered related to vaccination | Day 1 through Day 113
  According to the Medical Dictionary for Regulatory Activities (MedDRA) classification
Number of subjects reporting severe (Grade 3) laboratory Adverse Events (AE) considered related to vaccination | Day 1 through Day 92
  According to the Medical Dictionary for Regulatory Activities (MedDRA) classification
Number of subjects reporting solicited local reactions | Day 1 through Day 92
Number of subjects reporting solicited systemic reactions | Day 1 through Day 92
Number of subjects reporting unsolicited adverse events (AEs) considered related to vaccination and that are severe (Grade 3) | Day 1 through Day 113
  According to the Medical Dictionary for Regulatory Activities (MedDRA) classification

SECONDARY OUTCOMES:
Antibody titer against the malaria circumsporozoite antigen | Day 1 through Day 574
  Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Presence of P. falciparum asexual parasitemia following experimental malaria challenge | Day 118 to Day 141
Time to P. falciparum asexual parasitemia following experimental malaria challenge | Day 118 to Day 141

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Friedman-Klabanoff DJ, Berry AA, Travassos MA, Shriver M, Cox C, Butts J, Lundeen JS, Strauss KA, Joshi S, Shrestha B, Mo AX, Nomicos EYH, Deye GA, Regules JA, Bergmann-Leitner ES, Pasetti MF, Laurens MB. Recombinant Full-length Plasmodium falciparum Circumsporozoite Protein-Based Vaccine Adjuvanted With Glucopyranosyl Lipid A-Liposome Quillaja saponaria 21: Results of Phase 1 Testing With Malaria Challenge. J Infect Dis. 2024 Jun 14;229(6):1883-1893. doi: 10.1093/infdis/jiae062. PMID 38330357
- [Derived] Friedman-Klabanoff DJ, Berry AA, Travassos MA, Cox C, Zhou Y, Mo AX, Nomicos EYH, Deye GA, Pasetti MF, Laurens MB. Low dose recombinant full-length circumsporozoite protein-based Plasmodium falciparum vaccine is well-tolerated and highly immunogenic in phase 1 first-in-human clinical testing. Vaccine. 2021 Feb 22;39(8):1195-1200. doi: 10.1016/j.vaccine.2020.12.023. Epub 2021 Jan 22. PMID 33494963